CLINICAL TRIAL: NCT04792645
Title: A Double-Blind, Placebo-Controlled Study of Memantine in Body Focused Repetitive Behaviors
Brief Title: Memantine in Body Focused Repetitive Behaviors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB20-1992
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-07

CONDITIONS: Trichotillomania (Hair-Pulling Disorder); Dermatillomania
MeSH Terms: conditions — Trichotillomania; Excoriation Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 10mg once daily of placebo for two weeks, then 20mg for the remaining six weeks
  Interventions: Drug: Placebo
- Memantine (Experimental): 10mg once daily of memantine for two weeks, then 20mg for the remaining six weeks
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Placebo — Pill that contains no medicine
  Other Names: no other name
  Arms: Placebo
Drug: Memantine — Cognition-enhancing medication
  Other Names: Namenda
  Arms: Memantine

SUMMARY:
This study is 8 weeks long and involves subjects taking memantine or placebo. If they are randomly assigned to the memantine arm and are eligible to participate in the study, they will begin by taking 10mg once daily of memantine for two weeks, then 20mg for the remaining six weeks. Efficacy and safety measures will be performed at each visit. Participants will be randomized to receive either memantine or placebo on a 1:1 basis. This blinding will be maintained by the IDS pharmacy at the University of Chicago.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of memantine in 100 subjects with DSM-5 trichotillomania (TTM) or skin picking disorder (SPD).

The hypothesis to be tested is that memantine will be more effective and well tolerated in adults with trichotillomania or skin picking disorder compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder where there are not any current treatments options.

This will be one of few studies assessing the use of pharmacotherapy for the treatment of TTM and SPD in adults. Assessing the efficacy and safety of memantine will help inform clinicians about additional treatment options for adults suffering from this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age ≥18 years;
2. current DSM-5 trichotillomania or skin picking disorder; and
3. Ability to understand and sign the consent form.

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
4. Past 12-month DSM-5 diagnosis of psychosis, bipolar disorder, mania, or a substance or alcohol use disorder
5. Illegal substance use based on urine toxicology screening
6. Stable dose of medications for at least the past 3 months
7. Previous treatment with memantine
8. Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant JE, Chamberlain SR. Trichotillomania. Am J Psychiatry. 2016 Sep 1;173(9):868-74. doi: 10.1176/appi.ajp.2016.15111432. PMID 27581696
- [Background] Grant JE, Odlaug BL, Chamberlain SR, Keuthen NJ, Lochner C, Stein DJ. Skin picking disorder. Am J Psychiatry. 2012 Nov;169(11):1143-9. doi: 10.1176/appi.ajp.2012.12040508. PMID 23128921
- [Background] Grant JE, Odlaug BL, Hampshire A, Schreiber LR, Chamberlain SR. White matter abnormalities in skin picking disorder: a diffusion tensor imaging study. Neuropsychopharmacology. 2013 Apr;38(5):763-9. doi: 10.1038/npp.2012.241. Epub 2012 Nov 29. PMID 23303052
- [Background] Grant JE, Chamberlain SR, Redden SA, Leppink EW, Odlaug BL, Kim SW. N-Acetylcysteine in the Treatment of Excoriation Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):490-6. doi: 10.1001/jamapsychiatry.2016.0060. PMID 27007062
- [Background] Grant JE, Odlaug BL, Chamberlain SR, Kim SW. A double-blind, placebo-controlled trial of lamotrigine for pathological skin picking: treatment efficacy and neurocognitive predictors of response. J Clin Psychopharmacol. 2010 Aug;30(4):396-403. doi: 10.1097/JCP.0b013e3181e617a1. PMID 20531220
- [Background] Cloninger CR, Przybeck TR, Svrakic DM. The Tridimensional Personality Questionnaire: U.S. normative data. Psychol Rep. 1991 Dec;69(3 Pt 1):1047-57. doi: 10.2466/pr0.1991.69.3.1047. PMID 1784653

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Memantine
Started | 45 | 55
Completed | 36 | 43
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine | Total
Number analyzed (Participants) | 45 | 55 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.82 (11.46) | 30.25 (9.08) | 31.41 (10.25)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 33 | 47 | 80
  Gender: Male | 9 | 6 | 15
  Gender: Other Gender | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 39 | 44 | 83
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 55 | 100
National Institute of Mental Health Trichotillomania Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The National Institute of Mental Health Trichotillomania Symptom Severity Scale (NIMH-TTM) is a standard clinician administered scale to assess trichotillomania symptom severity. Scale range of 0-20. Higher scores indicate greater severity.
  units on a scale | 12.02 (3.30) | 12.67 (3.21) | 12.34 (3.23)
Massachusetts General Hospital Hairpulling Scale [Mean (Standard Deviation); unit: units on a scale] — A standard self-report scale to assess trichotillomania symptom severity. Scale ranges 0-28. Higher scores indicate greater severity.
  units on a scale | 19.57 (3.52) | 19.30 (4.41) | 19.42 (4.01)
Sheehan Disability Scale [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) is a self-report measure designed to assess functional impairment. Participants indicate how much their symptoms have disrupted their work/school, social life, and family/home responsibilities. Score ranges from 0-30, with higher scores indicating greater functional impairment.
  units on a scale | 9.43 (7.75) | 10.23 (7.19) | 9.87 (7.44)
HAM-A [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Scale (HAM-A) is a clinician-rated scale used to assess level of anxiety in participants. Score ranges from 0-56, with higher scores indicating greater anxiety.
  units on a scale | 5.20 (5.67) | 6.89 (5.55) | 6.13 (5.60)
HAM-D [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale (HAM-D) is a clinician-rated self-report measure designed to assess for depression symptoms in participants. Scores range from 0-58, with higher scores indicating more depression symptoms.
  units on a scale | 4.29 (3.80) | 5.87 (4.12) | 5.16 (3.98)

OUTCOME MEASURES:

1. Primary Outcome: NIMH Symptom Severity Scale (for TTM or Skin Picking)
Description: The primary efficacy measure will be the change in hair pulling or skin picking frequency and urges to pull hair or pick skin for the past week as indicated by change in total score. The entire study lasts 10 weeks. Every two weeks subjects will take the NIMH Symptom Severity Scale. The change in scores from baseline to after 8 weeks will be assessed. The scale itself assesses severity of trichotillomania or skin picking symptom, with higher scores indicating greater trichotillomania or skin picking severity. Score range: 0-20.
Time Frame: The primary efficacy end points will be the change in these measures from baseline to week 8.
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 36 | 43
units on a scale | -1.19 (2.80) | -6.98 (3.65)

2. Secondary Outcome: Clinical Global Impressions-Improvement Scale (CGI-I)
Description: The entire study for the subject will last 8 weeks. Every two weeks the subject will complete the CGI-I. The scale is a clinician-rated measure of overall disorder severity. Scores range from 1 (not at all improved) to 7 (very much improved). In each group, the number of people in each group who had a CGI-I score of 6 or 7 at Week 8 (indicating much or very much improved) will be presented.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 36 | 43
participants | 3 | 26

3. Secondary Outcome: Massachusetts General Hospital Hairpulling (Skin Picking) Scale
Description: Brief, self-report scale for assessing repetitive hairpulling (or skin picking). Because of a lack of an identical scale for skin-picking behavior, this scale was modified for skin picking for individuals with SPD to keep the outcome measure consistent across disorders. Seven individual items, rated for severity from 0 to 4, assess urges to pull (pick), actual pulling (picking), perceived control, and associated distress (range 0-28). The change in scores from baseline to after 8 weeks is reported. Negative values indicate a decrease in score from baseline to 8 weeks, while positive values indicate an increase in score from baseline to 8 weeks.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 36 | 43
units on a scale | -3.09 (4.43) | -6.95 (4.20)

4. Secondary Outcome: Skin Picking Symptom Assessment Scale
Description: The entire study lasts 8 weeks. Every two weeks subjects will take the Skin Picking Symptom Assessment Scale (SP-SAS). The scale itself assesses severity of skin-picking symptoms. The SP-SAS score ranges from 0 to 48, with 0 being no symptoms and 48 being the most severe. The average change in score from baseline to Week 8 will be reported for both groups. A positive value indicates an increase in score from baseline to week 8, whereas a negative value indicates a decrease in score from baseline to week 8.
Time Frame: 8 weeks
Population: This assessment was only completed for participants with a diagnosis of skin picking disorder, even though the study was open to people who had either trichotillomania or skin picking disorder. This is why the sample size is smaller for analysis of this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 16 | 19
units on a scale | -2.44 (4.50) | -7.00 (8.74)

5. Secondary Outcome: Sheehan Disability Scale
Description: Subjects will complete the Sheehan Disability Scale (SDS) at all visits. The SDS is a self-report measure of functional impairment. Scores range from 0-30, with higher scores indicating greater functional impairment. The average change in score from baseline to Week 8 will be reported. Negative values indicate a decrease in score from baseline to Week 8, while positive values indicate an increase in score.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 36 | 43
units on a scale | -1.66 (7.25) | -5.73 (5.76)

6. Secondary Outcome: Hamilton Depression Rating Scale
Description: A clinician-administered assessment of depression that will be assessed at all study visits. Score range 0-58. Higher total scores indicate higher levels of depression, while a score of 0 would indicate no depressive symptoms. The change in score from baseline to Week 8 is reported. Positive values indicate an increase in score from baseline to Week 8, whereas negative values indicate a decrease in score from baseline to Week 8.
Time Frame: 8 weeks
Population: Participants who had HAM-D data at Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 36 | 42
units on a scale | -1.31 (3.95) | -2.90 (3.57)

7. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: A clinician-administered assessment of anxiety that will be assessed at all study visits. Score range: 0-56. Higher scores indicate more anxiety symptoms, with 0 being no symptoms of anxiety. Changes in scores from baseline to week 8 visit will be assessed. Positive values indicate an increase in score from baseline to week 8, whereas negative values indicate a decrease in score from baseline to week 8.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 36 | 43
units on a scale | -1.42 (5.20) | -3.88 (4.89)

8. Secondary Outcome: Quality of Life Inventory (QOLI)
Description: The entire study for an individual subject will last 8 weeks. This inventory will be completed at the first and last visit of the study, with only these two points being assessed. Results are reported as the change in Week 8-Week 0 scores. The scale itself assess the subjects overall perceived quality of life, with higher scores indicating better outcomes. Possible total scores range from 1-77.
Time Frame: 8 weeks
Population: Participants who had QOLI data at Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 37 | 32
units on a scale | 2.76 (19.87) | -0.09 (11.27)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 10-week study period .
Arm/Group | Placebo | Memantine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/55
Other Adverse Events (participants affected / at risk) | 13/45 | 15/55
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | Memantine (N=55)
Fatigue (General disorders) | 4 (5) | 4 (5)
Dizziness (General disorders) | 2 (3) | 4 (4)
Brain Fog (Nervous system disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (4)
Dry Mouth (General disorders) | 3 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Insomnia (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04792645/Prot_SAP_001.pdf